CLINICAL TRIAL: NCT03116685
Title: A Phase III Double-blind, Randomised Study to Evaluate the Long-term Efficacy and Safety of Oxabact in Patients With Primary Hyperoxaluria
Brief Title: A Study to Evaluate the Efficacy and Safety of Oxabact in Patients With Primary Hyperoxaluria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OxThera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC5-DB-02
Record Dates: First submitted 2017-04-07; First posted 2017-04-17 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-10

CONDITIONS: Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria, Primary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxabact OC5 capsules (Experimental): Oxabact OC5 - Oxalobacter formigenes HC-1
  Interventions: Biological: Oxabact OC5 - Oxalobacter formigenes HC-1
- Placebo capsules (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Oxabact OC5 - Oxalobacter formigenes HC-1 — Active study drug
  Arms: Oxabact OC5 capsules
Other: Placebo — Placebo
  Arms: Placebo capsules

SUMMARY:
This study will evaluate the efficacy and safety of OC5 in patients with PH.

DETAILED DESCRIPTION:
To evaluate the efficacy of Oxabact following 52 weeks treatment in subjects with maintained kidney function, but below the lower limit of the normal range (estimated glomerular filtration rate [eGFR] < 90 ml/min/1.73 m2) and a total plasma oxalate (Pox) concentration ≥ 10 μmol/L. Parameters to be evaluated include the ability to stabilise/reduce Pox concentration, to stabilise/improve kidney function and to reduce oxalate deposits in primary hyperoxaluria (PH) subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (as applicable for the age of the subject)
2. A diagnosis of PH (as determined by standard diagnostic methods).
3. eGFR < 90 ml/min/1.73 m2. The Schwartz formula will be used to estimate GFR for children (age below 18), and CKD-EPI formula will be used for adults (age 18 or above).
4. Plasma oxalate concentration ≥10 μmol/L in total plasma oxalate.
5. Male or female patients ≥ 2 years of age.
6. Patients receiving vitamin B6 must be receiving a stable dose for at least 3 months prior to screening and must not change the dose during the study. Patients not receiving vitamin B6 at study entry must be willing to refrain from initiating pyridoxine during study participation.

Exclusion Criteria:

1. Inability to swallow size 4 capsules.
2. Subjects that have undergone transplantation (solid organ or bone marrow).
3. Patients requiring dialysis or at immediate risk for kidney failure or expected to be in need of dialysis during the study period.
4. The existence of secondary hyperoxaluria, e.g. hyperoxaluria due to bariatric surgery or chronic gastrointestinal diseases such as cystic fibrosis, chronic inflammatory bowel disease and short-bowel syndrome.
5. Use of antibiotics to which O. formigenes is sensitive. (This includes current antibiotic use, or antibiotics use within 14 days of initiating study medication).
6. Current treatment with a separate ascorbic acid preparation.
7. Pregnant women (or women who are planning to become pregnant) or lactating women.
8. Women of childbearing potential who are not using adequate contraceptive precautions. Please see section 7.3 regarding requirements for contraception.
9. Presence of a medical condition that the Investigator considers likely to make the subject susceptible to adverse effect of study treatment or unable to follow study procedures or any condition that is likely to interfere with the study drug mechanism of action (such as abnormal GI function).
10. Participation in any interventional study of another investigational product, biologic, device, or other agent within 60 days prior to the first dose of OC5 or not willing to forego other forms of investigational treatment during this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gesa Schalk, MD, Principal Investigator — KindernierenZentrum, Bonn, Germany
Locations (10):
- Vanderbilt University Hospital, Nashville, Tennessee, United States
- Centre Hospitalier Universitaire de Liège, Liège, Belgium
- Hôpital Robert Debré, Paris, France
- Kindernierenzentrum Bonn, Bonn, Germany
- Hospital Vall d' Hebron, Barcelona, Spain
- Tunisia (3):
  - Hédi Chaker University Hospital, Sfax
  - Sahloul University Hospital, Sousse
  - Charles Nicolle University Hospital, Tunis
- United Kingdom (2):
  - Royal Free Hospital, London
  - Nottingham Children's Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 09 January 2018. Primary study completion 15 April 2021
Period: Overall Study
Arm/Group | Oxabact OC5 Capsules | Placebo Capsules
Started | 13 | 12
Completed | 13 | 11
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxabact OC5 Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 8 | 18
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (6.4) | 18.3 (16.5) | 15.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 2 | 3
  United States | 0 | 1 | 1
  United Kingdom | 1 | 2 | 3
  Tunisia | 3 | 1 | 4
  Germany | 2 | 4 | 6
  Spain | 6 | 2 | 8
Primary Hyperoxaluria Type [Count of Participants; unit: Participants] — Primary Hyperoxaluria is the result of rare genetic mutations. The three main types of primary hyperoxaluria are the result of different gene deficiencies.
  Primary Hyperoxaluria Type I is the result of mutations in the AGXT gene (alanine-glyoxylate aminotransferase) Primary Hyperoxaluria Type II is the result of mutations in the GRHPR gene (glyoxylate reductase-hydroxypyruvate reductase)
  Participants
    PH Type I | 13 | 11 | 24
    PH Type II | 0 | 1 | 1
Stage of Chronic Kidney Disease [Count of Participants; unit: Participants] — Chronic Kidney Disease is categorized in five stages: I-V based on kidney function.
  Stage I is mild damage with an eGFR of 90 or greater Stage II is mild damage with an eGFR between 60 and 89 Stage III is moderate damage with an eGFR between 30 and 59
  Participants
    Stage I | 1 | 2 | 3
    Stage II | 11 | 5 | 16
    Stage III | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Oxalate Concentration After 52 Weeks of Treatment
Description: Change from baseline in total plasma oxalate concentration after 52 weeks of treatment in micromole/liter
Time Frame: 52 weeks
Population: Full analysis set using a mixed repeated measures model for change for missing data
Measure: Mean (Standard Deviation); unit: micromole/liter
Arm/Group | Oxabact OC5 Capsules | Placebo Capsules
Number analyzed (Participants) | 13 | 12
micromole/liter
  Baseline value | 14.8 (5.7) | 14.4 (5.4)
  Change from baseline to 52 weeks | -0.71 (1.34) | 2.35 (1.46)

2. Secondary Outcome: Change From Baseline in Kidney Function
Description: Evaluation based on eGFR calculation using the 2009 creatinine-based "Schwartz bedside" equation (for children below 18 years of age) (Schwartz et al., 2009) and 2009 creatinine-based CKD-EPI equation for adults (Levey et al., 2009). Subjects who turn 18 during the study period were continuously evaluated using the Schwartz equation, ie the equation used at baseline was kept throughout the study.
Time Frame: 52 weeks
Population: Patients with baseline and week 52 assessments
Measure: Least Squares Mean (Standard Error); unit: millilitres/minute/1.73m2
Arm/Group | Oxabact OC5 Capsules | Placebo Capsules
Number analyzed (Participants) | 12 | 8
millilitres/minute/1.73m2 | -1.35 (2.68) | -0.06 (3.12)

3. Secondary Outcome: Frequency of Kidney Stone Events
Description: Number of kidney stone events for each patient
Time Frame: Through week 48
Population: Number of events
Measure: Number; unit: Number of kidney stone events
Arm/Group | Oxabact OC5 Capsules | Placebo Capsules
Number analyzed (Participants) | 13 | 12
Number of kidney stone events | 7 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 52 week study period
Arm/Group | Oxabact OC5 Capsules | Placebo Capsules
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/13 | 4/12
Other Adverse Events (participants affected / at risk) | 13/13 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxabact OC5 Capsules (N=13) | Placebo Capsules (N=12)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (2) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxabact OC5 Capsules (N=13) | Placebo Capsules (N=12)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tact infection (Infections and infestations) | 1 (1) | 2 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal colic (Renal and urinary disorders) | 2 (7) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator may not publish the results of their cohort of subjects until the full study has been submitted for publication. They may not submit for publication or present the results of this study without allowing OxThera 30 days in which to review and comment on the pre-publication manuscript. The investigator may not submit the results of the study for publication without the prior consent of OxThera, unless the review period has passed and there has been no reaction from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03116685/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03116685/SAP_001.pdf